CLINICAL TRIAL: NCT02862015
Title: A Multicenter, Prospective, Randomized Clinical Trial of the Clinical Effectiveness of Oncothermia Combined With Standard Chemotherapy in Metastatic Pancreatic Cancer Patients
Brief Title: Multicenter RCT of the Clinical Effectiveness of Oncothermia With Chemotherapy in Metastatic Pancreatic Cancer Patients
Acronym: Oncothermia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hospicare Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-IMGPB-2016-03
Record Dates: First submitted 2016-08-07; First posted 2016-08-10 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Cancer, Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oncothermia (Experimental): Patients with oncothermia treatment and palliative chemotherapy
  Interventions: Other: Oncothermia; Drug: FOLFIRINOX or Gemcitabine based chemotherapy
- Control (Active Comparator): Patients with palliative chemotherapy only
  Interventions: Drug: FOLFIRINOX or Gemcitabine based chemotherapy

INTERVENTIONS:
Other: Oncothermia — Oncothermia is a kind of hyperthermia treatment. It serves heat energy more selectively than conventional hyperthermia.
  Arms: Oncothermia
Drug: FOLFIRINOX or Gemcitabine based chemotherapy — As a standard palliative chemotherapy, FOLFIRINOX or Gemcitabine based chemotherapy will be treated to the patients.

SUMMARY:
Patients with pancreatic cancer often suffer from pain. Because of such a pain, their quality of life have seriously deteriorated. There have been a few studies that showed an effect for pain control by hyperthermia (heating the patient's body). However, there are several limitations in conventional hyperthermia.

In a previous pilot study (NCT02150135), we found the improvement of quality of life, function, and symptom.

From this background, the investigators tried to show the effect of "Oncothermia" with conventional chemotherapy for pain control, increasing quality of life, and anti-tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed pancreatic adenocarcinoma
* Patients with radiologically identified metastasis (CT or MRI)
* Patients with no history of previous chemotherapy
* Patients with ECOG score 0-2

Exclusion Criteria:

* Patients who have an experience of hyperthermia treatment
* Patients who have a difficulty of sensing heat
* Patients who have a skin graft or breast reconstruction surgery
* Patients who have a cardiac pacemaker or an implanted metal
* Pregnant or breast feeding women
* Patients with uncontrolled infection, diabetes, hypertension, ischemic heart disease, myocardial infarct within 6 months
* Patients who were treated with unproved drugs within 30 days
* Patients who have a serious disease which can affect the person's safety
* Patients who do not consent to the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ)-C30 score change | 3 months

SECONDARY OUTCOMES:
change of opioid use amount | 3 months
change of pain score (VAS score) | 3 months
Adverse effect | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hyeok Hwang, MD PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No